CLINICAL TRIAL: NCT07393113
Title: CLarifying ABCB1's Role in Amyloid Efflux and Alzheimer's Disease Risk
Brief Title: CLarifying ABCB1's Role in Alzheimer's Disease
Acronym: CLeAR-AD
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251732
Record Dates: First submitted 2026-01-19; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; P-glycoprotein
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA samples stored in a biobank from patients followed in a memory clinic who underwent a lumbar puncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cerebrospinal fluid amyloid and phosphorylated tau biomarkers (A+T+)
  Interventions: Genetic: ABCB1 genotyping
- Patients without cerebrospinal fluid amyloid, phosphorylated tau and total tau biomarkers (A-T-N-)
  Interventions: Genetic: ABCB1 genotyping

INTERVENTIONS:
Genetic: ABCB1 genotyping — Genotyping of three single nucleotide polymorphisms (3435C>T, 2677G>T/A, and 1236C>T) associated with variation in P-glycoprotein activity, using DNA samples stored in a biobank.

SUMMARY:
Alzheimer's disease is biologically defined by the accumulation of amyloid beta and tau protein, identified using cerebrospinal fluid biomarkers. The ABCB1 gene, which encodes P-glycoprotein involved in amyloid beta efflux across the blood-brain barrier, may influence Alzheimer's disease risk. We hypothesize that certain functional ABCB1 polymorphisms impair amyloid beta clearance, thereby promoting the development of biologically defined Alzheimer's disease.

DETAILED DESCRIPTION:
A case-control study comparing the distribution of three functional ABCB1 gene polymorphisms (3435C>T, 2677G>T/A, 1236C>T) in patients with biologically defined Alzheimer's disease versus neurological controls. We will also analyze the distribution of haplotypes derived from the combination of these three polymorphisms and investigate potential interactions between these polymorphisms and the APOE genotype, particularly the presence of the ε4 allele.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 50 years,
* available cerebrospinal fluid biomarker results,
* an available and usable DNA sample,
* and consent for future research use within the biobank.

Exclusion Criteria:

* the presence of an active non-degenerative neurological disorder (for example, multiple sclerosis, infections, or tumors),
* and missing data regarding APOE genotyping or cardiovascular risk factors

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in a memory clinic who underwent a comprehensive clinical and paraclinical assessment, including cerebrospinal fluid biomarkers.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Allele and genotype frequencies of ABCB1 single nucleotide polymorphisms (3435C>T, 2677G>T/A, and 1236C>T) | Baseline (at the time of biological sampling and clinical assessment)
  Allele and genotype frequencies of the ABCB1 single nucleotide polymorphisms 3435C>T, 2677G>T/A, and 1236C>T, determined by genotyping from genomic DNA, will be compared between:
  * patients with biologically defined Alzheimer's disease (A+T+Nx), and
  * neurological control participants with a negative biomarker profile (A-T-N-). Data will be summarized as allele frequencies and genotype distributions in each group.

SECONDARY OUTCOMES:
Haplotype frequencies of ABCB1 polymorphisms (3435C>T, 2677G>T/A, and 1236C>T) | Baseline (at the time of biological sampling and clinical assessment)
  Haplotype frequencies derived from the combination of the ABCB1 single nucleotide polymorphisms 3435C>T, 2677G>T/A, and 1236C>T, inferred from genotyping data, will be compared between:
  * patients with biologically defined Alzheimer's disease (A+T+Nx), and
  * neurological control participants with a negative biomarker profile (A-T-N-). Haplotypes will be summarized as frequency distributions within each group.
Distribution of ABCB1 polymorphisms stratified by APOE ε4 carrier status | Baseline (at the time of biological sampling and clinical assessment)
  The distribution of ABCB1 single nucleotide polymorphisms (3435C>T, 2677G>T/A, and 1236C>T) will be assessed according to APOE ε4 carrier status (ε4 carriers vs non-carriers) in:
  * patients with biologically defined Alzheimer's disease (A+T+Nx), and
  * neurological control participants with a negative biomarker profile (A-T-N-). ABCB1 allele and genotype frequencies will be summarized within each APOE ε4 stratum.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lariboisière - Fernand Widal (AP - HP), Paris, France

IPD SHARING:
Plan to Share IPD: No